CLINICAL TRIAL: NCT04701684
Title: WE-TRUST (Workflow Optimization to Reduce Time to Endovascular Reperfusion for Ultra-fast Stroke Treatment)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: XCY607-130512
Record Dates: First submitted 2020-12-21; First posted 2021-01-08 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Direct tot Angiography Suite (DTAS) triage workflow (Experimental)
  Interventions: Device: Direct to Angio Suite (DTAS) Philips' CBCT triage
- Conventional CT/MR triage workflow (Active Comparator)
  Interventions: Procedure: Conventional CT/MR triage

INTERVENTIONS:
Device: Direct to Angio Suite (DTAS) Philips' CBCT triage — Stroke patients are diagnosed and treated (mechanical thrombectomy) in the same angio suite
  Arms: Direct tot Angiography Suite (DTAS) triage workflow
Procedure: Conventional CT/MR triage — First a CT or MRI exam is acquired for triage. In case of an ischemic stroke the patient is then treated in an interventional suite.
  Arms: Conventional CT/MR triage workflow

SUMMARY:
The WE-TRUST study is a multi-center randomized clinical trial to assess the impact of a Direct to Angio Suite (DTAS) workflow on stroke patient outcomes.

DETAILED DESCRIPTION:
Outcomes for stroke patients are closely tied to how fast they receive treatment. Currently, when a possible stroke patient arrives at the emergency department, typically first a CT or MRI exam is acquired for stroke triage. In case of an ischemic stroke the patient is then treated in an interventional suite.

In the DTAS workflow stroke patients are diagnosed and treated in the interventional suite without interruption. The Cone-Beam CT (CBCT) capabilities of the interventional X-ray system are utilized to perform triage, directly followed by stroke treatment.

The primary objective of the WE-TRUST study is to demonstrate that the DTAS triage workflow involving CBCT results in superior patient outcome in ischemic stroke patients with confirmed Large Vessel Occlusion as compared to the conventional CT/MR triage workflow.

The WE-TRUST study will be running in 16+ sites to enroll 500+ patients globally.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or older, or of legal age to give informed consent per state or national law.
* Baseline NIHSS score obtained prior to randomization must be equal or higher than 10 points.
* Subjects with no significant pre-stroke functional disability (modified Rankin scale 0 - 2).
* Subjects suspected of acute ischemic stroke with an estimated arrival time at a stroke center (clinical investigational site participating in this study) < 6 hours from symptom onset OR wake-up stroke with time last known well of < 12 hours and symptoms discovered within 6 hours from arrival time at a stroke center. Symptom onset is defined as point in time the patient was last known well (at baseline).
* Informed consent obtained from patient or his or her legally designated representative (if locally required).
* Angiography suite immediately available.
* Endovascular treatment team immediately available (Neurologist, Neurointerventionalist, Anesthesiologist, Nursing, Technicians as per local standard practice)

Exclusion Criteria:

Clinical exclusion criteria:

* Known hemorrhagic diathesis, coagulation factor deficiency, or oral anticoagulant therapy with INR > 3.0
* Known baseline platelet count < 30.000/μL
* Baseline blood glucose of < 50mg/dL (< 2.78mmol/l)
* For patients receiving thrombolysis: severe, sustained hypertension (SBP > 185 mm Hg or DBP > 110 mm Hg). Note: If the blood pressure can be successfully reduced and maintained at the acceptable level using AHA/ASA guidelines recommended medication (including IV antihypertensive drips), the patient can be enrolled.
* Patients from a transfer center (Primary Stroke Center) with a CT/MR that is not required to be redone in the Comprehensive Stroke Center as per discretion of the physician or per local standards (e.g. CT/MR less than 90 minutes old).
* Patients in coma (NIHSS item of consciousness >1) defined as totally unresponsive; responding only with reflexes or being areflexic (Intubated patients for transfer could be randomized only in case an NIHSS is obtained by a neurologist prior transportation).
* Patients with extreme vomiting
* Patients that are extremely agitated
* Seizures at stroke onset which would preclude obtaining a baseline NIHSS
* Serious, advanced, or terminal illness with anticipated life expectancy of less than one year.
* Patients acquired stroke while in-hospital
* History of life-threatening allergy (more than rash) to contrast medium
* Cerebral vasculitis
* Patients with a pre-existing neurological or psychiatric disease that would confound the neurological or functional evaluations, mRS score at baseline must be ≤2. This excludes patients who are severely demented, require constant assistance in a nursing home type setting or who live at home but are not fully independent in activities of daily living (toileting, dressing, eating, cooking and preparing meals, etc.)
* Unlikely to be available for 90-day follow-up (e.g. no fixed home address, visitor from overseas).
* Patients with unstable clinical status who require emergent life support care
* Any condition that, in the judgment of the investigator could impose hazards to the patient if study therapy is initiated or affect the participation of the patient in the study.
* Subject participates in a potentially confounding drug or device trial during the course of the study.
* Woman of childbearing potential who is known to be pregnant on admission.
* Subject meets an exclusion criteria according to national law (e.g. age, pregnant woman, breast feeding woman)
* Subject is Philips employee or their family members residing with this Philips employee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 594 (Estimated)
Dates: Start 2021-06-23 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Distribution of ordinal modified Rankin Scale (mRS) scores at 90 ± 14 days follow-up | 90 ± 14 days follow-up
  The difference in the distribution of ordinal modified Rankin Scale (mRS) scores at 90 ± 14 days follow-up in the Target population to determine the performance of the DTAS triage imaging workflow involving Stroke CBCT reconstructions by the investigational device or SmartCT R3 in comparison to the conventional CT/MR triage imaging workflow. The 90 day mRS score will be evaluated by a blinded assessor of a pool of blinded assessors (i.e., a specialist with mRS certification) at the local hospital by performing a structured interview of the patient in person using the Rankin Focused Assessment (RFA) structured mRS questionnaire. If the subject is unable to return to the clinic for the day 90 ± 14 visit, a (video) call in which the mRS score is assessed by a blinded assessor is preferable to no assessment.

SECONDARY OUTCOMES:
Median time measurements (door-to-arterial puncture time) | Peri-procedural time
  Door-to-arterial puncture time: Time patient arrives at the Comprehensive Stroke Center door to the time the skin of the patient is touched to perform first arterial puncture.
Median time measurements (door-to-reperfusion time) | Peri-procedural time
  Door-to-reperfusion time: Time patient arrives at the Comprehensive Stroke Center door to the time of successful vessel recanalization (eTICI ≥ 2b)
Distribution of ordinal modified Rankin Scale (mRS) scores | 90 ± 14 days follow-up
  The distribution of ordinal modified Rankin Scale (mRS) scores at 90 ± 14 days follow-up in both arms in the Randomized population.

OTHER OUTCOMES:
Safety: Adverse events (mortality at 90 days) | At 90 days post-procedure
  Mortality and stroke-related mortality
Safety: Adverse events (symptomatic ICH) | At 24 (-12/+24) hours
  All intracranial hemorrhages will be classified by the blinded Core Lab using the Heidelberg Bleeding Classification. Symptomatic ICH will be defined as per a modified SITS-MOST definition [31]: Symptomatic intracranial hemorrhage is defined as local or remote parenchymal hemorrhage type 2, subarachnoid hemorrhage, and/or intraventricular hemorrhage on the 24 (-12/+24) hours post-treatment imaging scan, combined with a neurological deterioration of 4 points or more on the NIHSS from baseline, or from the lowest NIHSS value between baseline and 24 (-12/+24) hours after randomization, or leading to death.
Safety: Adverse events (asymptomatic ICH) | At 24 (-12/+24) hours
  All intracranial hemorrhages will be classified (blinded) by using the Heidelberg Bleeding Classification. All the intracranial hemorrhages which are not symptomatic, are classified as asymptomatic.
Safety: Adverse events (other) | From start of enrollment until hospital discharge (e.g. up to 5 days)
  including information of the seriousness, treatment needed, resolution and relevant judgment concerning the causal relationship with the investigational device, SmartCT R3, comparator (CT/MR), or procedure will be summarized for safety information.
Safety: Adverse Device Effects | From start of enrollment until hospital discharge (e.g. up to 5 days)
  including information of the seriousness, treatment needed, resolution and relevant judgment concerning the causal relationship with the investigational devices, released SmartCT R3 product or procedure will be summarized for safety information.
Safety: Number of participants with Device Deficiencies that could have led to Serious Adverse Event | From start of enrollment until hospital discharge (e.g. up to 5 days)
  including any corrective actions taken during the study, if any, will be summarized for safety information.
Exploratory: Median time measurements (door-to-randomization time) | Peri-procedural time
  Door-to-randomization time: Time patient arrives at the Comprehensive Stroke Center door to the time of randomization
Exploratory: Median time measurements (door-to-imaging time) | Peri-procedural time
  Door-to-imaging time: Time patient arrives at the Comprehensive Stroke Center door to the time of initial triage imaging acquisition (i.e. non-contrast CBCT or CT/MR)
Exploratory: Median time measurements (randomization-to-imaging time) | Peri-procedural time
  Randomization-to-imaging time: Time of randomization to the time of initial triage imaging acquisition (i.e. non-contrast CBCT or CT/MR)
Exploratory: Median time measurements (randomization-to-puncture time) | Peri-procedural time
  Randomization-to-puncture time: Time of randomization to the time the skin of the patient is touched to perform first arterial puncture
Exploratory: Median time measurements (door-to-thrombolytics administration time) | Peri-procedural time
  Door-to-thrombolytics administration time: Time patient arrives at the CSC door to the time of start of thrombolytics administration.
Exploratory: Median time measurements (onset-to-door time) | Peri-procedural time
  Onset-to-door time: Time patient last seen well to the time the patient arrives at the Comprehensive Stroke Center door
Exploratory: Median time measurements (onset-to-arterial puncture time) | Peri-procedural time
  Onset-to-arterial puncture time: Time patient last seen well to the time the skin of the patient is touched to perform first arterial puncture
Exploratory: Median time measurements (onset-to-successful reperfusion (eTICI ≥ 2b) time) | Peri-procedural time
  Onset-to-successful reperfusion (eTICI ≥ 2b) time: Time patient last seen well to the time of successful vessel recanalization (based on angiogram).
Exploratory: Median time measurements (Emergency Medical Services call-to-door time) | Peri-procedural time
  Emergency Medical Services call-to-door time: Time from the call to Emergency Medical Services to the time the patient arrives at the Comprehensive Stroke Center door (total ambulance service time)
Exploratory: Median time measurements (Comprehensive Stroke Center notification call-to-door time) | Peri-procedural time
  Comprehensive Stroke Center notification call-to-door time: Time from notification call to the Comprehensive Stroke Center stroke team to the time the patient arrives at the Comprehensive Stroke Center door
Exploratory: Median time measurements (imaging-to-thrombolytics administration time) | Peri-procedural time
  Imaging-to-thrombolytics administration time: Time from initial triage imaging acquisition (i.e. non-contrast CBCT or CT/MR) to the time of start of thrombolytics administration.
Exploratory: Median time measurements (imaging-to-arterial puncture time) | Peri-procedural time
  Imaging-to-arterial puncture time: Time from initial triage imaging acquisition (i.e. non-contrast CBCT or CT/MR) to the time the skin of the patient is touched to perform first arterial puncture
Exploratory: Median time measurements (Door-to-device deployment (first pass) time) | Peri-procedural time
  Door-to-device deployment (first pass) time: Time patient arrives at the CSC door to the time of device deployment (first pass).
Exploratory: Median time measurements (imaging-to-successful reperfusion (eTICI ≥ 2b) time) | Peri-procedural time
  Imaging-to-successful reperfusion (eTICI ≥ 2b) time: Time from initial triage imaging acquisition (i.e. non-contrast CBCT or CT/MR) to time of successful vessel recanalization (based on angiogram).
Exploratory: Median time measurements (arterial puncture-to-successful reperfusion (eTICI ≥ 2b) time) | Peri-procedural time
  Arterial puncture-to-successful reperfusion (eTICI ≥ 2b) time: Time the skin of the patient is touched to perform first arterial puncture to the time of successful vessel recanalization.
Exploratory: Median time measurements (arterial puncture-to-end-of-EVT procedure (catheter out) time) | Peri-procedural time
  Arterial puncture-to-end-of-EVT procedure (catheter out) time: Time the skin of the patient is touched to perform first arterial puncture to the time of the catheter is taken out (total EVT procedure time)
Exploratory: Degree of disability (other clinical outcome) | At discharge or 5-7 days post-procedure, and at 90 ± 14 days post-procedure
  Defined as modified Rankin Scale score (scores 0-6) distribution at discharge or at 5-7 days post-procedure, whichever comes first, and at 90 ± 14 days.
Exploratory: NIHSS (other clinical outcome) | At admission (baseline), 24(-12/+24) hours after randomization, discharge or at 5-7 days post-procedure, whichever comes; and at 90 ± 14 days post-procedure
  The National Institutes of Health Stroke Scale is a tool used to objectively quantify the impairment caused by a stroke. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0
Exploratory: Functional independence (other clinical outcome) | At 90 ± 14 days post-procedure
  Functional independence defined as mRS ≤ 2 at 90 days. The scale runs from 0-6, running from perfect health without symptoms (0) to death (6).
Exploratory: UW-mRS (other clinical outcome) | At 90 ± 14 days post-procedure
  Utility-Weighted modified Ranking Scale. The scale runs from 0-6, running from perfect health without symptoms (0) to death (6).
Exploratory: Dichotomized mRS score (other clinical outcome) | At 90 ± 14 days post-procedure
  Dichotomized mRS score (0-3 versus 4-6). The scale runs from 0-6, running from perfect health without symptoms (0) to death (6).
Exploratory: Infarct volume (other clinical outcome) | At 24 (-12/+24) hours post-procedure
  Infarct volume evaluated on CT or MRI
Exploratory: Dramatic early favorable response (other clinical outcome) | At 24 (-12/+24) hours after randomization
  Defined as an NIHSS score of 0-2 or NIHSS improvement ≥ 8 points. The National Institutes of Health Stroke Scale is a tool used to objectively quantify the impairment caused by a stroke. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0
Exploratory: Successful vessel recanalization (other clinical outcome) | At the end of the endovascular procedure
  Defined as expanded Thrombolysis in Cerebral Infarction) (eTICI) grade 2b, 2c or 3 on the post-procedure angiogram
Exploratory: X-ray radiation exposure (other clinical outcome) | On day 1
  Total X-ray Radiation Exposure measured as effective dose (mSv).

CONTACTS AND LOCATIONS:
Overall Officials: Raul G Nogueira, Principal Investigator — UPMC Stroke Institute, Pittsburgh; Marc Ribo, Principal Investigator — Vall d'Hebron University Hospital, Barcelona
Locations (22):
- United States (3):
  - Baptist Medical Center, Jacksonville, Florida
  - Grady Memorial Hospital/Emory University, Atlanta, Georgia
  - Montefiore Medical Center, The Bronx, New York
- La Sagrada Familia Clinic, José Hernández, Argentina
- Brazil (3):
  - Hospital Geral de Fortaleza, Fortaleza
  - Hospital de Base, São José do Rio Preto
  - Hospital Estadual Central - Fundação Estadual de Inovação em Saúde - Inova Capixaba, Vitória
- France (3):
  - Hospices Civils de Lyon, Lyon
  - CHU Montpellier, Montpellier
  - Bicêtre Hospital, Paris
- Germany (4):
  - University Hospital Bonn (UKB Universitätsklinikum Bonn), Bonn
  - Klinikum Kassel, Kassel
  - Universitätsklinikum Schleswig-Holstein Lübeck, Lübeck
  - Klinikum rechts der Isar der TU München, Munich
- Netherlands (2):
  - St. Antonius Ziekenhuis, Nieuwegein
  - Haaglanden Medical Center, The Hague
- University Emergency Hospital Bucharest, Bucharest, Romania
- Spain (4):
  - Hospital Clinico San Carlos, Madrid, Moncloa - Aravaca
  - Vall d'Hebron University Hospital, Barcelona
  - Hospital Universitari Doctor Josep Trueta de Girona, Girona
  - Hospital Virgen del Rocio, Seville
- İstanbul Aydin University medical park florya hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: WE-TRUST study information website — https://www.wetrust-study.com/